CLINICAL TRIAL: NCT00330304
Title: Long Term Study of 2 Isoniazid (INH) Prophylactic Regimens With Concomitant Cotrimoxazole (CTX) in HIV-infected Children - Impact on Morbidity, Mortality, Bacterial Resistance and Incidence of Tuberculosis
Brief Title: Isoniazid Prophylaxis With Concomitant Cotrimoxazole in HIV-infected Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Stellenbosch (Other); Medical Research Council (Other Government); Rockefeller Foundation (Other)
Responsible Party: Principal Investigator, Heather Zar, Professor, University of Cape Town
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 299/2005
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Child; HIV; prophylaxis; mortality
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Trimethoprim, Sulfamethoxazole Drug Combination

ARMS (2):
- Isoniazid preventive therapy (Experimental): HIV infected children living in a high TB prevalence area receive isonaizid prophylaxis daily, together with cotrimoxazole prohpylaxis either 3 times a week or daily.
  Interventions: Drug: Isoniazid; Drug: Cotrimoxazole
- Placebo (Placebo Comparator): HIV infected children living in a high TB prevalence area receive placebo once daily
  Interventions: Drug: Cotrimoxazole; Other: placebo

INTERVENTIONS:
Drug: Isoniazid — isoniazid 10mg/kg orally, daily, for study period
  Arms: Isoniazid preventive therapy
Drug: Cotrimoxazole — Cotrimoxazole given 3 times a week or daily, orally, for study period
Drug: isoniazid — Isoniazid, 10mg/kg daily for study period
  Arms: Isoniazid preventive therapy
Other: placebo — Placebo tablet identicle in appearance to intervention: isoniazid table
  Arms: Placebo

SUMMARY:
The study involves use of isoniazid and cotrimoxazole as strategies for preventing infections in HIV-infected children and reducing mortality. Cotrimoxazole is well known to reduce mortality and infections in HIV-infected children and is currently the recommended standard of care. However, isoniazid has only been studied in HIV-infected adults (in whom it has been shown to substantially reduce the incidence of tuberculosis). In a randomised controlled study of isoniazid in HIV-infected children, the investigators found that INH reduced mortality and tuberculosis incidence in excess of 50%; the data safety monitoring board recommended termination of the placebo arm given the beneficial effects of INH. The investigators therefore aim to follow-up these children to compare the long term impact of two different INH and CTX preventive regimens (daily versus thrice weekly) on morbidity, mortality, adherence and incidence of adverse reactions. The investigators also aim to investigate the efficacy, safety and tolerability of INH compared with placebo for prevention of TB in children receiving HAART as the benefit in this group is unknown.

DETAILED DESCRIPTION:
Tuberculosis (TB) and HIV are dual pandemics occurring in South Africa. Prevention of TB and the subsequent decline in immune function in HIV-infected children is an important strategy to reduce mortality. Isoniazid (INH) prophylaxis reduces TB incidence in HIV-infected adults, but the efficacy in HIV-infected children has not been studied. In 2003, the investigators therefore began a double blind placebo controlled trial to investigate the impact of INH prophylaxis on mortality, morbidity and TB incidence in HIV-infected children. Interim analysis found a striking reduction in mortality and TB with a decrease in mortality in excess of 50% and 60% respectively, in children on INH. Based on this, the placebo arm was terminated; the study continued as a trial of thrice versus daily INH and cotrimoxazole (CTX). Although the results indicate an important benefit in children on INH, it is unknown what the long term efficacy and safety of INH prophylaxis is, what the optimal regime is and whether this pertains to children on HAART (who formed a minority of the cohort but who are still at risk for TB).

Aim To investigate the efficacy, safety and tolerability of INH and CTX as prophylactic strategies for HIV-infected children in a high TB prevalence area.

Objectives

1. To compare the long term impact of two different INH preventive regimens (daily versus thrice weekly) on TB incidence, occurrence of INH resistance in patients with culture-confirmed TB, mortality, incidence of adverse reactions and adherence
2. To compare the long term impact of two different CTX prophylactic regimens (daily versus thrice weekly) on mortality, frequency and duration of hospitalization, type of serious infections, nasopharyngeal carriage of bacteria and development of antimicrobial resistance, adherence and incidence of adverse reactions
3. To investigate the efficacy, safety and tolerability of INH compared with placebo for prevention of TB in children receiving HAART

Methods A prospective randomized double blind placebo controlled study of INH versus placebo in newly recruited HIV-infected children who are stable on HAART. In addition, an extended follow-up study of children already randomised to thrice weekly or daily INH and CTX. Children will be followed for 2 years with regular clinical evaluation, adherence assessment and laboratory monitoring. Outcomes measured will be mortality, TB incidence, morbidity, adherence and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children
* Resident in Cape Town
* Informed consent obtainable
* weight > 2.5kg
* Access to transport
* HAART use for not less than 2 months but not more than 12 months with no significant demonstrated toxicity and good adherence

Exclusion Criteria:

* Chronic diarrhoea
* Current use of INH prophylaxis
* Prior hypersensitivity to INH prior history of allergy to sulphur drugs
* Prior history of allergy to sulphur drugs
* Severe anaemia (haemoglobin less than 7 gm/dl)
* Neutropenia (absoloute neutrophil count less than 400 cells)
* Thrombocytopenia (platelet count < 50 000/uL)
* Non-reversible renal failure
* Clinical hepatitis
* Exposure to household TB contact, requiring INH prophylaxis

Ages: 8 Weeks to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2011-11-15 (Actual); Study Completion 2011-11-15 (Actual)

PRIMARY OUTCOMES:
TB incidence | Jan 2003 to July 2011
Mortality | Jan 2003 to July 2011

SECONDARY OUTCOMES:
intercurrent infections | Jan 2003 to July 2011
adherence | Jan 2003 to July 2011
adverse events | Jan 2003 to July 2011
antimicrobial resistance | Jan 2003 to July 2011

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Zar, MD PHd, Principal Investigator — University of Cape Town; Mark Cotton, Md PhD, Principal Investigator — University of Stellenbosch
Locations (2):
- South Africa (2):
  - Red Cross Childrens Hospital, Cape Town, Western Cape
  - Tygerberg Hospital, Cape Town, Western Cape

REFERENCES:
- [Derived] Amlabu V, Mulligan C, Jele N, Evans A, Gray D, Zar HJ, McIlleron H, Smith P. Isoniazid/acetylisoniazid urine concentrations: markers of adherence to isoniazid preventive therapy in children. Int J Tuberc Lung Dis. 2014 May;18(5):528-30. doi: 10.5588/ijtld.13.0730. PMID 24903787
- [Derived] Gray DM, Workman LJ, Lombard CJ, Jennings T, Innes S, Grobbelaar CJ, Cotton MF, Zar HJ. Isoniazid preventive therapy in HIV-infected children on antiretroviral therapy: a pilot study. Int J Tuberc Lung Dis. 2014 Mar;18(3):322-7. doi: 10.5588/ijtld.13.0354. PMID 24670570
- [Derived] Frigati LJ, Kranzer K, Cotton MF, Schaaf HS, Lombard CJ, Zar HJ. The impact of isoniazid preventive therapy and antiretroviral therapy on tuberculosis in children infected with HIV in a high tuberculosis incidence setting. Thorax. 2011 Jun;66(6):496-501. doi: 10.1136/thx.2010.156752. Epub 2011 Apr 2. PMID 21460373
- [Derived] le Roux SM, Cotton MF, Golub JE, le Roux DM, Workman L, Zar HJ. Adherence to isoniazid prophylaxis among HIV-infected children: a randomized controlled trial comparing two dosing schedules. BMC Med. 2009 Nov 3;7:67. doi: 10.1186/1741-7015-7-67. PMID 19886982
- [Derived] Zar HJ, Cotton MF, Strauss S, Karpakis J, Hussey G, Schaaf HS, Rabie H, Lombard CJ. Effect of isoniazid prophylaxis on mortality and incidence of tuberculosis in children with HIV: randomised controlled trial. BMJ. 2007 Jan 20;334(7585):136. doi: 10.1136/bmj.39000.486400.55. Epub 2006 Nov 3. PMID 17085459